CLINICAL TRIAL: NCT07202182
Title: The Effect of a Creative Drama-Based Stress Management Program on Stress, Coping, and Emotional Intelligence Levels in Nursing Students: A Single-Blind Randomized Controlled Study
Brief Title: Creative Drama-Based Stress Management Program on Stress, Coping, and Emotional Intelligence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sultan Ayaz Alkaya, Prof. Dr., Faculty of nursing, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2025-1375
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Perceived Stress; Coping Skills; Emotional Intelligence; Nursing Student
Keywords: Perceived Stress; Coping with Stress; Emotional Intelligence; nursing students

STUDY DESIGN:
Intervention Model Description: randomized trial with experimental and control groups
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Creative Drama Group (Experimental): A creative drama-based stress management program consisting of a total of 6 sessions, 3 weeks, will be applied to the experimental group.
  Interventions: Behavioral: Creative Drama-Based Stress Management Program
- Active Comparator Grup (Active Comparator): The active control group will be given 3 weeks of theoretical training.
  Interventions: Behavioral: Training

INTERVENTIONS:
Behavioral: Creative Drama-Based Stress Management Program — A creative drama-based stress management program is an intervention that aims to reduce nursing students' stress levels and increase their coping and emotional intelligence skills.
  Arms: Creative Drama Group
Behavioral: Training — In the study, the control group will receive training on a topic different from the experimental intervention for three weeks. This method aims to prevent any loss of motivation that might result from the control group not receiving any training. It also helps determine whether the effects observed in the experimental group are due solely to the creative drama-based stress management program or to the overall training process.
  Arms: Active Comparator Grup

SUMMARY:
The study was designed with a parallel-group randomized controlled experimental design to determine the effects of a creative drama-based stress management program on the stress, coping, and emotional intelligence levels of nursing students. Nursing students in the intervention group will receive a creative drama-based stress management program for a total of six sessions over three weeks. Students in the active control group will receive three weeks of theoretical training. Students will receive a posttest at the end of the intervention program (3 weeks), a first follow-up one month after the intervention, and a second follow-up three months later.

H0-1: There is no difference in perceived stress levels between the intervention group that underwent the creative drama intervention and the control group.

H0-2: There is no difference in biopsychosocial response levels between the intervention group that underwent the creative drama intervention and the control group.

H0-3: There is no difference in stress coping levels between the intervention group that underwent the creative drama initiative and the control group.

H0-4: There is no difference in emotional intelligence levels between the intervention group that underwent the creative drama initiative and the control group.

DETAILED DESCRIPTION:
Nursing students will be assigned to the intervention and control groups using a stratified, simple randomization method within the strata. Gender was taken into account to ensure homogeneity between groups. Students will be divided into two strata based on gender (male and female).

To prevent selection bias, data will be collected by an independent expert, and students will be assigned to the intervention and control groups using a randomization method. Participant numbers will be assigned to students when the preliminary assessment data is transferred to the computer. Student group assignment will be conducted by a biostatistician independent of the study.

To prevent reporting bias, the study data will be analyzed by a biostatistician. Because the interventions will be administered by the researcher, there will be no investigator blinding. Participant blinding will be achieved by administering the educational intervention to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Being a nursing student,
* Volunteering to participate in the study,
* Scoring high on the Perceived Stress Scale for Nursing Students

Exclusion Criteria:

* Taking a creative drama course,
* Receiving professional psychological support,
* Having an illness that would prevent participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale for Nursing Students | Pre-intervention (pre-test) Immediately after the intervention (post-test) 1 month after the intervention (1st follow-up) 3 months after the intervention (2nd follow-up)
  Developed in Chinese by Sheu et al. (2002), the Turkish adaptation was made by Karaca et al. (2015). The scale consists of 29 items, and a five-point Likert-type scale was used to evaluate the items: "4 - Very stressful for me, 3, 2, 1, 0 - Not stressful for me." The scale has six subscales. The total score ranges from 0 to 116. A higher score indicates a higher degree of stress.
Bio-Psycho-Social Response Scale for Nursing Students | Pre-intervention (pre-test) Immediately after the intervention (post-test) 1 month after the intervention (1st follow-up) 3 months after the intervention (2nd follow-up)
  Developed in Chinese by Sheu et al. (2002), the Turkish adaptation was made by Karaca et al. (2015). The scale consists of 21 items, and a five-point Likert-type rating scale was used for the assessment of items: 4 - I always experience, 3, 2, 1, and 0 - I never experience. The scale has three subscales. A higher score indicates more symptoms and a poorer bio-psycho-social status.
Stress Coping Behaviors Scale for Nursing Students | Pre-intervention (pre-test) Immediately after the intervention (post-test) 1 month after the intervention (1st follow-up) 3 months after the intervention (2nd follow-up)
  Developed in Chinese by Sheu et al. (2002) and adapted into Turkish by Karaca et al. (2015). The scale consists of 19 items and was evaluated using a five-point Likert-type scale (4 - Agree, 3, 2, 1, 0 - Strongly Disagree). The scale has four subscales. A higher score on each subscale indicates that the student used that coping strategy more frequently.
Emotional Intelligence Trait Scale - Short Form | Pre-intervention (pre-test) Immediately after the intervention (post-test) 1 month after the intervention (1st follow-up) 3 months after the intervention (2nd follow-up)
  Developed by Petrides and Furnham (2000) to assess an individual's self-perception of their emotional abilities. Adapted to Turkish by Deniz et al. (2013), the scale consists of a total of 20 items and four subscales: well-being, self-control, emotionality, and sociability. A high score indicates a high level of emotional intelligence; a low score indicates a low level of emotional intelligence.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No